CLINICAL TRIAL: NCT02133703
Title: Decision Making Interventions for Women Receiving Uninformative BRCA1/2 Test Results or Positive BRCA1/2 Test Results
Brief Title: Decision Support Following Genetic Testing for Breast-Ovarian Cancer Susceptibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010-611; R01CA135179-01 (NIH); R01HG005055 (NIH)
Record Dates: First submitted 2014-04-09; First posted 2014-05-08 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: Genetic counseling; genetic testing; BRCA1; BRCA2; Hereditary breast cancer; Hereditary ovarian cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Breast Cancer, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Mutation Carrier: Enhanced Internet DA (Experimental): BRCA1/2 carriers randomized to this arm will have access to Internet-based decision support including a preference clarification tool.
  Interventions: Behavioral: Enhanced Internet DA
- Mutation Carrier: Internet DA (Experimental): BRCA1/2 carriers randomized to this arm will have access to Internet-based decision support intervention without a preference clarification tool.
  Interventions: Behavioral: Internet DA
- Mutation Carrier: Enhanced Print DA (Active Comparator): BRCA1/2 carriers randomized to this arm will be sent a print-based decision aid with a print preference clarification tool.
  Interventions: Behavioral: Enhanced Print DA
- Mutation Carrier: Print DA (Active Comparator): BRCA1/2 carriers randomized to this arm will receive a print decision aid without a preference clarification tool.
  Interventions: Behavioral: Print DA
- Inconclusive Results: DA (Experimental): Participants who receive inconclusive results who are randomized to this arm will have access to an Internet decision tool designed to facilitate management decision making
  Interventions: Behavioral: Inconclusive Results DA
- Inconclusive Results: Usual care (No Intervention): Participants who receive inconclusive/uninformative results who are randomized to this arm will receive usual care but no additional decision support intervention

INTERVENTIONS:
Behavioral: Enhanced Internet DA — BRCA1/2 carriers randomized to this arm will have access to Internet-based decision support including a preference clarification tool. This intervention is designed to provide education and decision support regarding the available risk management options.
  Arms: Mutation Carrier: Enhanced Internet DA
Behavioral: Internet DA — BRCA1/2 carriers randomized to this arm will have access to Internet-based decision support. This intervention is designed to provide education regarding the available risk management options.
  Arms: Mutation Carrier: Internet DA
Behavioral: Enhanced Print DA — BRCA1/2 carriers randomized to this arm will receive print-based decision support materials which include a preference clarification tool. This intervention is designed to provide education and decision support regarding the available risk management options.
  Arms: Mutation Carrier: Enhanced Print DA
Behavioral: Print DA — BRCA1/2 carriers randomized to this arm will receive print education materials designed to provide information regarding the available risk management options.
  Arms: Mutation Carrier: Print DA
Behavioral: Inconclusive Results DA — Women who receive uninformative BRCA1/2 results randomized to this arm will have access to Internet-based decision support including a preference clarification tool. This intervention is designed to provide education and decision support regarding the available risk management options.
  Arms: Inconclusive Results: DA

SUMMARY:
This non-therapeutic trial is for women who have received results of genetic testing for BRCA1/2 mutations. The trial compares decision support tools designed to facilitate informed decision making regarding risk management following testing to usual care. The researchers will test separate decision support tools for women who receive positive test results and women who receive negative/inconclusive test results. Among women who receive a positive test result, an interactive decision support intervention will be compared to a print intervention. Among women who receive an inconclusive result, an interactive intervention will be compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Undergo BRCA1/2 genetic counseling and testing at one of four study sites
* Receive positive or uninformative test results
* English speaking

Exclusion Criteria:

* Newly diagnosed breast cancer patients who have not yet initiated definitive breast cancer treatment
* Previous bilateral mastectomy

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2015-10; Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Knowledge | 1-month post randomization
  Knowledge of risk management options.
Decision Conflict | 1-month post-randomization
  Decisional Conflict Scale
Decision Satisfaction | 12-months post-randomization
  Satisfaction with Decision Scale
Psychological Distress | 1-month post randomization
Health Related Quality of Life | 12-months post randomization
  SF-12
Utilization of breast and ovarian cancer risk management options | 12-months post-randomization
  We will assess uptake of the following risk management strategies:
  1. Risk reducing surgery (mastectomy and oophorectomy)
  2. Chemoprevention
  3. Breast and ovarian cancer screening

SECONDARY OUTCOMES:
Knowledge | 3-months post randomization
  Knowledge of risk management options
Psychological Distress | 3-months post-randomization
Decisional Conflict | 3-months post-randomization
  Decisional Conflict Scale

CONTACTS AND LOCATIONS:
Overall Officials: Marc D Schwartz, PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center/Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States